CLINICAL TRIAL: NCT00061724
Title: Medical and Surgical Treatment of Esophageal Reflux
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: MSTER (completed)
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Esophageal; Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this project is to lay the groundwork for a proposed clinical trial to compare the effectiveness of two approaches to gastroesophageal reflux disease: treatment with medications and treatment with anti-reflux surgery. This project includes a non-interventional pilot study to test ways of measuring outcomes of treatment, and to gauge potential participants' willingness to enroll in the proposed clinical trial.

ELIGIBILITY:
Inclusion criteria:

* age 18-80
* diagnosis of gastroesophageal reflux disease
* have taken proton pump inhibitor medications

Exclusion criteria:

* prior esophageal surgery
* other serious medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hines VA Medical Center, Maywood, Illinois
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina